CLINICAL TRIAL: NCT06435299
Title: Efficacy and Tolerance of Cannabidiol in Patients with Severe Pruritus: a Multicenter, Double-blind, Randomized, Placebo-controlled Study
Acronym: CANNABITCH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 29BRC23.0164
Record Dates: First submitted 2024-03-27; First posted 2024-05-30 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabis oil (Experimental): Cannabis oil 50mg/mL arm :
  An auto-titration phase will take place during the first 14 days of treatment: 0.2 ml on the first day then increase of 0.2 ml every 2 days in 2 daily doses, that is to say 1.4 ml/day maximum.
  If any tolerable side-effects occurred, patients were advised not to increase the dose; if intolerable side-effects occurred, dose reduction was advised.
  After initial titration, the dose will then be maintained for 4 consecutive weeks.
  Interventions: Drug: Cannabis oil
- PLACEBO (Placebo Comparator): Placebo arm :
  An auto-titration phase will take place during the first 14 days of treatment: 0.2 ml on the first day then increase of 0.2 ml every 2 days in 2 daily doses, that is to say 1.4 ml/day maximum.
  If any tolerable side-effects occurred, patients were advised not to increase the dose; if intolerable side-effects occurred, dose reduction was advised.
  After initial titration, the dose will then be maintained for 4 consecutive weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabis oil — Patients in this arm will have to take Cannabis oil (50mg/mL) twice a day with the daily dose estimated during auto titration phase (from W0 to W2)
  Arms: Cannabis oil
Drug: Placebo — Patients in this arm will have to take Placebo oil twice a day with the daily dose estimated during auto titration phase (from W0 to W2)
  Arms: PLACEBO

SUMMARY:
Pruritus is defined as an unpleasant sensation leading to the need to scratch. Medications for pruritus are much less effective than those used for pain and it is imperative to find new therapeutic options.

Over the last 20 years, the understanding of the pathophysiology of pruritus has progressed significantly, opening new possible therapeutic fields. Among these, cannabinoids seem very promising because the physiological inhibitory role of endocannabinoids, mainly produced by neurons, has been well demonstrated. Data from the literature suggest that the antipruritic effects of cannabinoids are due to a combination of effects on neuronal activation, transmission along the afferent pathway, and local modulation of keratinocytes and mast cells. The antipruritic effect is peripheral and central, through modulation of CB1, CB2 or TRPV1 channels. CB1 and CB2 receptors are specific cannabinoid receptors, CB1 being present at the central and peripheral level while CB2 is only peripheral and very present in the skin. Cannabinoids can also bind to TRPV1, and thus inhibit neurogenic inflammation by antagonizing or stabilizing this ion channel, which prevents neuronal activation by pruritogenic mediators. Phytocannabinoids are derived from cannabis and are used for a variety of purposes, with their development for medical purposes expanding rapidly. The two best known are tetrahydrocannabinol (THC) and cannabidiol (CBD). THC binds to TRPV1, CB2 and CB1, the activation of the latter being at the origin of parallel psychotropic effects. CBD binds mainly to TRPV1, which allows us to expect very favorable effects on pruritus, neurogenic inflammation and skin pain, without fearing side effects of this type.

A limited number of studies suggest that cannabinoids may be useful topically or systemically, in humans or animals, but no comparative study with placebo has been performed. These encouraging results have been observed in cases of induced pruritus, idiopathic pruritus, eczema, uremic pruritus, cholestatic pruritus, prurigo, sensitive skin or even epidermolysis bullosa.

Currently, the ANSM is conducting an evaluation of the effects of medical cannabis on severe pain. We propose to evaluate the effects on severe pruritus in a randomized placebo-controlled study one of the products chosen by the ANSM in this context, the oil LITTLE GREEN PHARMA, which we choose for its dominant CBD ratio (THC < 5 mg/ml, CBD > 5 mg/ml).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Severe pruritus, defined by a mean WI-NRS score ≥7/10 (evaluated on one week before inclusion, regardless of the cause of the pruritus
* Insufficient relief (WI-NRS ≥7/10 ) or poor tolerance (adverse effects) of accessible drug and non-drug therapies
* Stable treatment (for treatment of the prurit) for at least 6 weeks
* Affiliated or benefiting of a social security
* Informed consent (personally dated and) signed by the participant or any representatives (impartial witness/trusted person)

Exclusion Criteria:

* Patients unable to consent.
* Patients refusing to participate in research.
* Patients under guardianship or conservatorship.
* Personal history of psychotic disorders.
* Severe hepatic impairment, defined as prothrombin level <50% or with predictive biological impairment.
* Moderate to severe renal impairment, with an estimated glomerular filtration rate ≤ 44 mL/min/1.73 m².
* Severe cardiovascular or cerebrovascular disease, including history of myocardial infarction or stroke.
* Pregnant or breastfeeding women.
* Lack of understanding of questionnaires or inability to follow up.
* Women of childbearing potential unwilling to use appropriate contraception.
* Cannabinoid use outside the clinical trial
* Use of cannabis or its derivatives less than one week before inclusion
* History of hypersensitivity or allergy to any cannabinoid product.
* Allergy to nuts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
WI-NRS change | Week 0
  Binary outcome (success or failure). Success is defined by a reduction of 30% in WINRS (Worst Itching Intensity Numerical Rating Scale - On a scale of 0 (no itch) to 10 (worst itch imaginable)) from the inclusion visit to week 6.
WI-NRS change | Week 6
  Binary outcome (success or failure). Success is defined by a reduction of 30% in WINRS (Worst Itching Intensity Numerical Rating Scale - On a scale of 0 (no itch) to 10 (worst itch imaginable)) from the inclusion visit to week 6.

SECONDARY OUTCOMES:
WI-NRS change from W0 to W2 | Week 0
  - Proportion of patients achieving at least a weekly mean reduction of 4 points in WI-NRS (Worst Itching Intensity Numerical Rating Scale - On a scale of 0 (no itch) to 10 (worst itch imaginable)) score from inclusion visit to week 2
WI-NRS change from W0 to W2 | Week 2
  - Proportion of patients achieving at least a weekly mean reduction of 4 points in WI-NRS (Worst Itching Intensity Numerical Rating Scale - On a scale of 0 (no itch) to 10 (worst itch imaginable)) score from inclusion visit to week 2
WI-NRS change from W2 to W6 | Week 2
  Proportion of patients achieving at least a weekly mean reduction of 4 points in WI-NRS (Worst Itching Intensity Numerical Rating Scale - On a scale of 0 (no itch) to 10 (worst itch imaginable)) score from week 2 to week 6.
WI-NRS change from W2 to W6 | Week 6
  Proportion of patients achieving at least a weekly mean reduction of 4 points in WI-NRS (Worst Itching Intensity Numerical Rating Scale - On a scale of 0 (no itch) to 10 (worst itch imaginable)) score from week 2 to week 6.
ItchyQoL change from W0 to W2 | Week 0
  - Change in ItchyQoL score from inclusion (= Week 0) visit to week 2 (The ItchyQoL questionnaire contains 22 items, and each item is rated on a 5-point scale, ranging from 1 = never to 5 = all the time)
ItchyQoL change from W0 to W2 | Week 2
  - Change in ItchyQoL score from inclusion (= Week 0) visit to week 2 (The ItchyQoL questionnaire contains 22 items, and each item is rated on a 5-point scale, ranging from 1 = never to 5 = all the time)
ItchyQoL change from W2 to W6 | Week 2
  - Percent change in ItchyQoL score from Week 2 visit to week 6 (The ItchyQoL questionnaire contains 22 items, and each item is rated on a 5-point scale, ranging from 1 = never to 5 = all the time)
ItchyQoL change from W2 to W6 | Week 6
  - Change in ItchyQoL score from Week 2 visit to week 6.(The ItchyQoL questionnaire contains 22 items, and each item is rated on a 5-point scale, ranging from 1 = never to 5 = all the time)
Chronic Itch Burden Scale change from W0 to W2 | Week 0
  - Change in Chronic Itch Burden Scale - 10 from inclusion (= Week 0) visit to week 2 (10 questions rated from "Not at all" to "Very much" on patient itching)
Chronic Itch Burden Scale change from W0 to W2 | Week 2
  - Change in Chronic Itch Burden Scale - 10 from inclusion (= Week 0) visit to week 2 (10 questions rated from "Not at all" to "Very much" on patient itching)
Chronic Itch Burden Scale change from W2 to W6 | Week 2
  - Percent change in Chronic Itch Burden Scale - 10 from Week 2 visit to week 6 (10 questions rated from "Not at all" to "Very much" on patient itching)
Chronic Itch Burden Scale change from W2 to W6 | Week 6
  - Percent change in Chronic Itch Burden Scale - 10 from Week 2 visit to week 6 (10 questions rated from "Not at all" to "Very much" on patient itching)
Treatment adverse events | Week 0
  - Incidence and severity of treatment-emergent adverse events.
Treatment adverse events | Week 2
  - Incidence and severity of treatment-emergent adverse events.
Treatment adverse events | Week 4
  - Incidence and severity of treatment-emergent adverse events.
Treatment adverse events | Week 6
  - Incidence and severity of treatment-emergent adverse events.
Treatment adverse events | Week 8
  - Incidence and severity of treatment-emergent adverse events.
Treatment Observance Rate | Week 6
  - Number of observant patients (YES/NO) in both arms: Observance (defined as YES) is considered as taking at least one dose of treatment per day over the W0 - W6 period.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU Angers, Angers, France
  - CHD Vendée, La Roche-sur-Yon, France
  - Groupe Hospitalier La Rochelle, La Rochelle, France
  - CHU de Nantes, Nantes, France
  - CHU de Poitiers, Poitiers, France
  - CHU de Rennes, Rennes, France
  - CHRU de Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided